CLINICAL TRIAL: NCT00808379
Title: Concurrent Chemo-Radiotherapy vs Radiotherapy With Boost in Locally Advanced Unresectable Rectal Cancers. A Randomized Phase II Study
Brief Title: Concurrent Chemo-Radiotherapy Versus Radiotherapy With Boost in Locally Advanced Unresectable Rectal Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Dr Reena Engineer (Principal Investigator), Tata Memorial Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 260
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Rectal Cancer
Keywords: Unresectable rectal cancers
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 2 (Radiation + boost ) (Other): Radiation dose to pelvis will be delivered at 1.8 Gy per day, five days per week, to give a total of 25 fractions over a period of five weeks for a total of 45 Gy.
  Boost Field - Will be given to all the patients in the radiotherapy alone followed by surgery arm.
  The boost will be given with by 3dimensional conformal radiotherapy to a dose of 15-20 Gy. After 45Gy the boost will be planned on the original tumor volume.
  Interventions: Radiation: Additional Radiation boost to the primary tumor volume
- Arm 1 (standard) Chemoradiation (Active Comparator): The Radiation dose will be delivered at 1.8 Gy per day, five days per week, to give a total of 25 fractions over a period of five weeks for a total of 45 Gy.
  Chemotherapy will begin on the first day of radiotherapy and continue until the completion of radiotherapy. Capecitabine will be administered orally daily 2000 mg/m2 in two divided doses (approximately 12 hours apart) for 2 weeks followed by a 1-week rest period given as 3 week cycles.
  Interventions: Drug: Chemoradiation

INTERVENTIONS:
Drug: Chemoradiation — Chemotherapy will begin on the first day of radiotherapy and continue until the completion of radiotherapy. Capecitabine will be administered orally daily 2000 mg/m2 in two divided doses (approximately 12 hours apart) for 2 weeks followed by a 1-week rest period given as 3 week cycles.
  Other Names: Capebine
  Arms: Arm 1 (standard) Chemoradiation
Radiation: Additional Radiation boost to the primary tumor volume — 15-20Gy
  Other Names: Radiation Boost
  Arms: Arm 2 (Radiation + boost )

SUMMARY:
At Tata Memorial Hospital 50% of the patients present in the locally advanced stage which is technically unresectable, or that is beyond the realm of a potentially curative surgical resection. The evaluation of treatment approaches for these tumors is hampered by the absence of any substantial randomized studies and the heterogeneous nature of the tumors at presentation.

The management of these tumors has changed over the years, there is emphasis on neoadjuvant chemoradiation therapy, trying to convert a tumor that is initially unresectable to one that is potentially curable by surgery. But only 70-80% of the patients are able to complete this treatment without any significant treatment breaks.

Dose escalated treatment with radiotherapy in locally advanced and unresectable rectal cancers have been tried in many small series with good results and lesser toxicity.

Comparison outcome between the two arms will indicate the relative efficacy and toxicity of neoadjuvant concurrent chemoradiation vs boosted radiotherapy alone in downstaging of advanced cancers.

DETAILED DESCRIPTION:
Aims/ Objectives

1. To compare the resectability rate when patients are treated when conventional chemoradiation to patients treated with radiation alone with an additional boost to the primary tumor in case of unresectable rectal cancers.
2. To study the treatment toxicity and local control rate.

Study methodology This is a phase II Randomised controlled study. Ninety cases of advanced rectal cancer (Stage II - Stage III) will be divided in two equal groups (Arm I & II) Arm-1(standard arm) - Patients will receive standard external radiation therapy to pelvis + concurrent chemotherapy with Tab Capecitabine. This will be followed by surgery at 6-8 weeks if deemed resectable.

Arm-2 (research arm) Patients in this group will not receive any neo-adjuvant chemotherapy, instead they will receive radiotherapy alone additional dose of localized radiotherapy boost. This will be followed by surgery at 6-8 weeks if deemed resectable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable disease, medically able to undergo pelvic surgery.
2. Patients with unresectable adenocarcinoma of the rectum located up to 12 cm from the anal verge without evidence of distant metastases.
3. Patients must be 18 years old or greater.
4. Patients with clinical stage T3 orT4 based on endorectal ultrasound or physical exam.
5. Patients with lab values within standard protocol parameters
6. Karnofsky performance status > 60.
7. No history of other malignancies within 5 years, except non-melanoma skin cancer, in situ carcinoma of the cervix or ductal carcinoma of the breast. Previous invasive cancer permitted if disease-free at least 5 years
8. Patient must sign study-specific consent prior to randomization.

Exclusion Criteria:

1. Any evidence of distant metastasis
2. Synchronous primary colon carcinomas, except T1 lesions
3. Prior radiation therapy to the pelvis
4. Prior chemotherapy for malignancies
5. Pregnancy or lactation.
6. Serious, uncontrolled, concurrent infection(s).
7. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
8. Evidence of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
9. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
10. Major surgery within 4 weeks of the study treatment.
11. Lack of physical integrity of the upper gastrointestinal tract or mal-absorption syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of resectability rate of in the two groups at 6-8 weeks following radiotherapy. | 3 years
Side effects and other adverse effects in the two groups during radiotherapy and up to 2 years post radiotherapy. | 3 years

SECONDARY OUTCOMES:
Comparison of pathological downstaging between the two groups who undergo surgery. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Reena Engineer, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India